CLINICAL TRIAL: NCT03193658
Title: Effect of Ultrasound Guided Bilateral Thoracolumbar Interfascial Plane (TLIP) Block on Post-operative Opioid Consumption After Lumbar Spine Surgeries. A Randomized Double Blinded Study.
Brief Title: USG Thoracolumbar Interfascial Plane (TLIP) in Lumbar Spine Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eslam Ayman Mohamed Shawki (Other)
Responsible Party: Sponsor-Investigator, Eslam Ayman Mohamed Shawki, Lecturer of anesthesia, SICU & Pain Management, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: TLIP_spine
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Regional Anesthesia
Keywords: spine surgery; Thoracolumbar Interfascial Plane block; regional anesthesia; postoperative analgesia; opioid consumption
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: Randomized controlled double blinded study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T (Active Comparator): Will receive bilateral US guided Thoracolumbar Interfascial Plane (TLIP) block at the proposed level of surgery before the start of the surgery
  Interventions: Procedure: Thoracolumbar Interfascial Plane (TLIP) block
- Group O (Active Comparator): Will not receive the block and postoperative pain control will be managed by I.V drug based multi-modal approach (Opioid & acetaminophen) only.
  Interventions: Drug: I.V drug based multimodal approach

INTERVENTIONS:
Procedure: Thoracolumbar Interfascial Plane (TLIP) block — A 10 cm 21G Stimuplex needle (Braun Medical Inc, Bethlehem, PA, USA) will be inserted in a lateral-to-medial orientation with an approximate angle of 30 degrees to the skin. The needle will then be advanced under real-time in-plane ultrasound guidance through the belly of the LG towards the MF. The needle tip will be directed towards the LG/MF interface deep to the midpoint then a total volume of 20 ml of Bupivacaine 0.25% will be incrementally injected with intermittently repeated negative aspiration. Anterior spread of local anesthetic will be viewed as favourable.
  The same procedure will be repeated on the left side. The patient will then be disinfected and draped and surgery will be allowed to proceed normally.
  Arms: Group T
Drug: I.V drug based multimodal approach — A base low dose opioid of 5mg morphine I.V every 8 hours. Rescue analgesia will be given to the patient if reported a VAS equal or more than 4 in the form of I.V morphine in 2.5mg increments till VAS returns to 4 or less in addition to 1 gm of oral acetaminophen every 6 hours
  Arms: Group O

SUMMARY:
The study aims to evaluate the effect of US guided bilateral Thoracolumbar Interfascial plane (TLIP) block performed at the level of the lumbar spine surgery (involving 1 up to 3 adjacent lumbar vertebrae) after induction of general anesthesia and before starting the surgery on postoperative opioid consumption by the patients during the first 24 hours postoperative.

DETAILED DESCRIPTION:
Commonly performed spinal surgeries include laminectomies and discectomies, spinal fusions, and instrumentations, scoliosis corrections and spinal tumor excision. Conventional non-minimally invasive spinal surgeries usually involve extensive dissection of subcutaneous tissues, bones, and ligaments and thus can result in a considerable degree of postoperative pain. The severe pain typically last for at least 3 days with the highest pain scores recorded during the first 24 hours postoperative. Pain from the back originates from different tissues such as vertebrae & intervertebral discs, facet joint capsules, dura & nerve root sleeves, ligaments, fascia, and muscles, and it is directly proportional to the number of vertebrae involved in the surgery. Sensations from these structures are carried via the posterior rami of spinal nerves connected to sympathetic & parasympathetic nerves.

Adequate pain management in this period can result in improved functional outcome, early ambulation, early discharge, and preventing the development of chronic pain. Many options exist for this purpose, but each has its limitations and applications. The postoperative multi-modal analgesic approach to these patients include drugs like NSAIDs, acetaminophen, opioids, gabapentinoids and even corticosteroids, but using drugs alone for pain management in these patients can prove to be problematic due to side effects like GIT problems (NSAIDs), urinary retention, respiratory depression , nausea & vomiting (opioids), in addition, prescribing postoperative opioids will be more complicated if the patient was on prolonged preoperative opioid regimen (due to the associated opioid resistance), that's why patients on opioids prior to surgery reported more time postoperatively spent in severe pain (60% versus 38%; p=-0.002).

Multiple loco-regional techniques were explored to help supplement the multi-modal approach to decrease side effects, improve quality of postoperative analgesia, increase patient satisfaction after lumbar spine surgeries and also to be used in Enhanced Recovery After Surgery (ERAS) protocols which aims at minimizing opioid analgesics whenever possible. Via-Catheter techniques considered include patient-controlled epidural analgesia that showed promising results regarding pain control but concerns were raised due to its interference with postoperative assessment of neurological functions & voiding, in addition, it was opposed by many surgeons due to the fact of putting a catheter very near to the surgical field. Also continuous infusion of local anesthetics was explored which resulted in decreased postoperative opioid consumption but also raised concerns due to the catheter being placed very near to the wound.

Single injection methods that were explored in the literature include local anesthetic instillation of the affected nerve roots by the surgeon before wound closure, wound local anesthetic infiltration, and even a single low dose of intrathecal morphine administered by the surgeon into the intrathecal space under direct visualization at the conclusion of the surgery. But none of these methods was widely accepted due to limitations in the duration and adequacy of postoperative analgesia.

US guided Thoracolumbar Interfascial plane (TLIP) block is a novel technique first described in a pilot study on volunteers published by William R. Hand and colleagues in Nov 2015, it was designed to target the dorsal rami of the thoracolumbar nerves as they pass through the paraspinal musculature (between the multifidus muscle (MF) and the longissimus muscle (LG)), which is analogous to the Transversus Abdominis plane (TAP) block which targets the ventral rami of the thoracolumbar nerves (between the Transversus Abdominis muscle and the internal oblique muscle).

The block was performed bilaterally at the level of L3 and they reported a reproducible area of anesthesia to pinprick in a mean (SD) area covering 137.4 (71.0) cm2 of the lower back (including the midline) after 20 minutes of the block.

Multiple case reports for TLIP block in lumbar spine surgery were described afterwards, Hironobu Ueshima and colleagues described 2 cases that required no additional postoperative analgesia and no complications, then another 2 cases with nearly the same results, they conducted a cadaveric study to assess the spread of injectate within the plane between the MF and LG muscles using only 5ml of blue dye solution, they verified the spread of the dye to the transverse process of the 3rd lumbar vertebra (level of injection) in all cadavers, so they suggested that the local anesthetic's injectate into the fascial plane between the MF and LG muscles can indeed block the posterior rami of the lumbar nerves.

Finally they explored the continuous variation of the block in another 2 cases with reported pain free duration for 2 days (the duration of the study) and a pinprick anesthesia area covering from L1 to L4 level and no complications.

TLIP block has the potential benefit of blocking sensations from spinal and para-spinal structures involved in the surgical trauma up to 1 level above and below the level of the block (including deeper structures, not only skin and subcutaneous tissues, unlike simple wound infiltration), while also sparing neurological functions of the lower limb (specially the motor functions) and urinary bladder functions (Voiding).

ELIGIBILITY:
Inclusion Criteria:

- Adult patients undergoing lumbar spine surgeries involving 1 up to 3 adjacent lumbar vertebrae (eg. laminectomy, discectomy …).

Exclusion Criteria:

* Patients on preoperative opioid regimen for more than 1 month.
* Patients with history of previous surgical operations in the lumbar region.
* Patients with spinal deformities (eg. Scoliosis…..).
* Hypersensitivity to Bupivacaine.
* Extensive Lumbar spine surgeries like large tumour excisions, scoliosis correction or more than 2 level spine fixation.
* Patients with communication difficulties.
* Lumbar spine operations that will be performed with the patient in any position other than the prone position.
* Severe neurological compromise (severe muscle weakness such as foot drop or sphincter disorders such as urinary incontinence).
* Coagulopathies with prothrombin concentration less than 60% or INR more than 1.5.
* In-ability to postpone anti-coagulation medications.
* Infection, injury or a lesion at the block site.
* ASA class 3 and 4 patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption in the first 24 hours postoperative | 24 hours postoperative
  Total morphine consumption in the first 24 hours postoperative (Above the basal 15mg given to all patients) as an indicator of technique efficiency in improving postoperative analgesia.

SECONDARY OUTCOMES:
Time required to perform the technique | 30 minutes
  Time required to perform the technique (time between the start of US scanning and injection of the second local anesthetic bolus).
Time of the operation | 4 hours
  Time of the operation (time between induction of anesthesia and full recovery of the patient)
Total intraoperative I.V. fentanyl dose | 4 hours
  Total intraoperative I.V. fentanyl dose (above the standard 2µg/kg).
VAS value after recovery | 4 hours
  VAS value obtained from patient immediately after recovery from anesthesia then every 4 hours during the first 24 hours postoperatively.
Modified Bromage score value after recovery | 4 hours
  Modified Bromage score value in the lower limbs obtained immediately after recovery from anesthesia then every 4 hours during the first 24 hours postoperatively.
First time of rescue analgesia | 24 hours
  First time of rescue analgesia
Incidence of side effects related to opioid use | 24 hours
  Incidence of side effects related to opioid use (postoperative nausea and vomiting (PONV), constipation, pruritus, urinary retention…..).
Incidence of complications or side-effects related to the block | 24 hours
  Incidence of complications or side-effects related to the block (hematoma formation or intravascular injection).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Cairo University teaching hospitals (Kasr Alainy), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bianconi M, Ferraro L, Ricci R, Zanoli G, Antonelli T, Giulia B, Guberti A, Massari L. The pharmacokinetics and efficacy of ropivacaine continuous wound instillation after spine fusion surgery. Anesth Analg. 2004 Jan;98(1):166-172. doi: 10.1213/01.ANE.0000093310.47375.44. PMID 14693613
- [Background] Klimek M, Ubben JF, Ammann J, Borner U, Klein J, Verbrugge SJ. Pain in neurosurgically treated patients: a prospective observational study. J Neurosurg. 2006 Mar;104(3):350-9. doi: 10.3171/jns.2006.104.3.350. PMID 16572646
- [Background] Bajwa SJ, Haldar R. Pain management following spinal surgeries: An appraisal of the available options. J Craniovertebr Junction Spine. 2015 Jul-Sep;6(3):105-10. doi: 10.4103/0974-8237.161589. PMID 26288544
- [Background] Devin CJ, McGirt MJ. Best evidence in multimodal pain management in spine surgery and means of assessing postoperative pain and functional outcomes. J Clin Neurosci. 2015 Jun;22(6):930-8. doi: 10.1016/j.jocn.2015.01.003. Epub 2015 Mar 9. PMID 25766366
- [Background] Aminmansour B, Khalili HA, Ahmadi J, Nourian M. Effect of high-dose intravenous dexamethasone on postlumbar discectomy pain. Spine (Phila Pa 1976). 2006 Oct 1;31(21):2415-7. doi: 10.1097/01.brs.0000238668.49035.19. PMID 17023848
- [Background] Tan M, Law LS, Gan TJ. Optimizing pain management to facilitate Enhanced Recovery After Surgery pathways. Can J Anaesth. 2015 Feb;62(2):203-18. doi: 10.1007/s12630-014-0275-x. Epub 2014 Dec 10. PMID 25501696
- [Background] Schenk MR, Putzier M, Kugler B, Tohtz S, Voigt K, Schink T, Kox WJ, Spies C, Volk T. Postoperative analgesia after major spine surgery: patient-controlled epidural analgesia versus patient-controlled intravenous analgesia. Anesth Analg. 2006 Nov;103(5):1311-7. doi: 10.1213/01.ane/0000247966.49492.72. PMID 17056975
- [Background] Reynolds RA, Legakis JE, Tweedie J, Chung Y, Ren EJ, Bevier PA, Thomas RL, Thomas ST. Postoperative pain management after spinal fusion surgery: an analysis of the efficacy of continuous infusion of local anesthetics. Global Spine J. 2013 Mar;3(1):7-14. doi: 10.1055/s-0033-1337119. Epub 2013 Mar 2. PMID 24436846
- [Background] Gurbet A, Bekar A, Bilgin H, Korfali G, Yilmazlar S, Tercan M. Pre-emptive infiltration of levobupivacaine is superior to at-closure administration in lumbar laminectomy patients. Eur Spine J. 2008 Sep;17(9):1237-41. doi: 10.1007/s00586-008-0676-z. Epub 2008 Apr 19. PMID 18425538
- [Background] Hand WR, Taylor JM, Harvey NR, Epperson TI, Gunselman RJ, Bolin ED, Whiteley J. Thoracolumbar interfascial plane (TLIP) block: a pilot study in volunteers. Can J Anaesth. 2015 Nov;62(11):1196-200. doi: 10.1007/s12630-015-0431-y. Epub 2015 Jul 7. PMID 26149600
- [Background] Kjaergaard M, Moiniche S, Olsen KS. Wound infiltration with local anesthetics for post-operative pain relief in lumbar spine surgery: a systematic review. Acta Anaesthesiol Scand. 2012 Mar;56(3):282-90. doi: 10.1111/j.1399-6576.2011.02629.x. Epub 2012 Jan 19. PMID 22260370
- [Background] Kumar A, Sinha C, Kumar A, Bhadani UK. Ultrasound-guided thoracolumbar interfascial plane block for spine surgery. Saudi J Anaesth. 2017 Apr-Jun;11(2):248-249. doi: 10.4103/1658-354X.203052. No abstract available. PMID 28442976
- [Background] Ueshima H, Oku K, Otake H. Ultrasound-guided thoracolumbar interfascial plane block: a cadaveric study of the spread of injectate. J Clin Anesth. 2016 Nov;34:259-60. doi: 10.1016/j.jclinane.2016.04.060. Epub 2016 May 13. No abstract available. PMID 27687388 (Retraction: PMID 35393195 J Clin Anesth. 2022 Aug;79:110771)
- [Background] Ueshima H, Hiroshi O. RETRACTED: Clinical experiences of the continuous thoracolumbar interfascial plane (TLIP) block. J Clin Anesth. 2016 Nov;34:555-556. doi: 10.1016/j.jclinane.2016.06.004. Epub 2016 Jul 19. No abstract available. PMID 27687450 (Retraction: PMID 35461753 J Clin Anesth. 2022 Aug;79:110737)
- [Background] Breen TW, Shapiro T, Glass B, Foster-Payne D, Oriol NE. Epidural anesthesia for labor in an ambulatory patient. Anesth Analg. 1993 Nov;77(5):919-24. doi: 10.1213/00000539-199311000-00008. PMID 8214727